CLINICAL TRIAL: NCT06315881
Title: Informing Oral Nicotine Pouch Regulations to Promote Public Health
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brittney Keller-Hamilton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-23116; NCI-2024-00666 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U54CA287392 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-03-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Specimen Handling; Tobacco Products; Tobacco, Smokeless

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- PHASE I ARM I (low FBN R/S ONP) (Experimental): Participants insert low free-base nicotine (FBN) R/S ONP product over 30 minutes and insert usual brand of ST over 30 minutes or smoke usual brand of cigarette over 5 minutes during each study visit for 5 visits over up to 3 months. Patients also undergo blood sample collection throughout study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration
- PHASE I ARM II (low FBN > 99% S ONP) (Experimental): Participants insert low FBN > 99% S ONP product over 30 minutes and insert usual brand of ST over 30 minutes or smoke usual brand of cigarette over 5 minutes during each study visit for 5 visits over up to 3 months. Patients also undergo blood sample collection throughout study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration
- PHASE I ARM III (high FBN R/S ONP) (Experimental): Participants insert high R/S ONP product over 30 minutes and insert usual brand of ST over 30 minutes or smoke usual brand of cigarette over 5 minutes during each study visit for 5 visits over up to 3 months. Patients also undergo blood sample collection throughout study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration
- PHASE I ARM IV (high FBN > 99% ONP) (Experimental): Participants insert high FBN > 99% S ONP product over 30 minutes and insert usual brand of ST over 30 minutes or smoke usual brand of cigarette over 5 minutes during each study visit for 5 visits over up to 3 months. Patients also undergo blood sample collection throughout study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration
- PHASE I ARM V (Usual brand ST or cigarette) (Experimental): Participants insert usual brand of ST over 30 minutes or smoke usual brand of cigarette over 5 minutes. Patients also undergo blood sample collection at 0, 5, 15, 30, 60, and 90 minutes.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Smokeless Tobacco; Other: Survey Administration
- PHASE II ARM I (low FBN R/S ONP) (Experimental): WASHOUT PERIOD: Participants use usual brand of ST or cigarettes for 1 week.
  CONTROL WEEK: Participants continue regular use of ST or cigarettes for 1 week and receive a text with a link to daily diary surveys to record tobacco use.
  Participants insert low FBN R/S ONP for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration; Other: Text Message-Based Navigation Intervention
- PHASE II ARM II (low FBN > 99% S ONP) (Experimental): WASHOUT PERIOD: Participants use usual brand of ST or cigarettes for 1 week.
  CONTROL WEEK: Participants continue regular use of ST or cigarettes for 1 week and receive a text with a link to daily diary surveys to record tobacco use.
  Participants insert to low FBN > 99% S ONP product for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration; Other: Text Message-Based Navigation Intervention
- PHASE II ARM III (high R/S ONP) (Experimental): WASHOUT PERIOD: Participants use usual brand of ST or cigarettes for 1 week.
  CONTROL WEEK: Participants continue regular use of ST or cigarettes for 1 week and receive a text with a link to daily diary surveys to record tobacco use.
  Participants insert to high R/S ONP product for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration; Other: Text Message-Based Navigation Intervention
- PHASE II ARM IV (high FBN > 99% ONP) (Experimental): WASHOUT PERIOD: Participants use usual brand of ST or cigarettes for 1 week.
  CONTROL WEEK: Participants continue regular use of ST or cigarettes for 1 week and receive a text with a link to daily diary surveys to record tobacco use.
  Participants insert high FBN > 99% S ONP product for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.
  Interventions: Procedure: Biospecimen Collection; Drug: Cigarette; Drug: Nicotine Oral Pouch; Drug: Smokeless Tobacco; Other: Survey Administration; Other: Text Message-Based Navigation Intervention

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample and oral mucosa sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cigarette — Smoke usual brand cigarette
Drug: Nicotine Oral Pouch — Insert low FBN R/S ONP
  Other Names: ZYN
  Arms: PHASE I ARM I (low FBN R/S ONP); PHASE II ARM I (low FBN R/S ONP)
Drug: Nicotine Oral Pouch — Insert low FBN > 99% S ONP
  Other Names: ZYN
  Arms: PHASE I ARM II (low FBN > 99% S ONP); PHASE II ARM II (low FBN > 99% S ONP)
Drug: Nicotine Oral Pouch — Insert high R/S ONP
  Other Names: ZYN
  Arms: PHASE I ARM III (high FBN R/S ONP); PHASE II ARM III (high R/S ONP)
Drug: Nicotine Oral Pouch — Insert high FBN > 99% ONP
  Other Names: ZYN
  Arms: PHASE I ARM IV (high FBN > 99% ONP); PHASE II ARM IV (high FBN > 99% ONP)
Drug: Smokeless Tobacco — Insert ST
  Other Names: Smoking, Tobacco and Cancer - Smokeless Tobacco
Other: Survey Administration — Ancillary studies
Other: Text Message-Based Navigation Intervention — Receive text with a link to daily diary surveys
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: PHASE II ARM I (low FBN R/S ONP); PHASE II ARM II (low FBN > 99% S ONP); PHASE II ARM III (high R/S ONP); PHASE II ARM IV (high FBN > 99% ONP)

SUMMARY:
This clinical trial evaluates the characteristics of oral nicotine pouches (ONPs) to determine if they are a comparable substitute to cigarette or smokeless tobacco (ST) products. ONPs contain nicotine but no tobacco and are used primarily by adult tobacco uses in the United States (US). ONPs are recognized by the Food and Drug Administration as having lower risk than combustible cigarettes and are approved as a modified risk tobacco product. While ONPs have lower toxic risk than other tobacco products, acute and longer term harm related to their use has not been studied. Information gathered from this study may identify product characteristics of ONPs that improve successful switching from high-risk cigarettes or ST to lower risk ONPs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the effects of nicotine concentration, form, and isomer on the satisfaction and appeal of ONPs relative to cigarettes and ST.

II. Evaluate the effects of nicotine concentration, form, and isomer on switching from cigarettes or ST to ONPs.

EXPLORATORY OBJECTIVE:

I. Examine changes in oral microbiome-host interactions associated with degree of switching from cigarettes/ST to ONPs.

OUTLINE:

PHASE I: Participants are randomized to use one of the 4 study ONP products or their usual product brand of ST or cigarette in either the low or high nicotine concentration arm.

ARM I: Participants insert low free-base nicotine (FBN) R/S ONP product over 30 minutes. Patients also undergo blood sample collection at 0, 5, 15, 30, 60, and 90 minutes.

ARM II: Participants insert low FBN > 99% S ONP product over 30 minutes. Patients also undergo blood sample collection at 0, 5, 15, 30, 60, and 90 minutes.

ARM III: Participants insert high R/S ONP product over 30 minutes. Patients also undergo blood sample collection at 0, 5, 15, 30, 60, and 90 minutes.

ARM IV: Participants insert high FBN > 99% S ONP product over 30 minutes. Patients also undergo blood sample collection at 0, 5, 15, 30, 60, and 90 minutes.

ARM V: Participants insert usual brand of ST over 30 minutes or smoke usual brand of cigarette over 5 minutes. Patients also undergo blood sample collection at 0, 5, 15, 30, 60, and 90 minutes.

PHASE II:

WASHOUT PERIOD: Participants use usual brand of ST or cigarettes for 1 week.

CONTROL WEEK: Participants continue regular use of ST or cigarettes for 1 week and receive a text with a link to daily diary surveys to record tobacco use.

PHASE II SWITCH: Participants are randomized to switch to 1 of 4 study ONP.

ARM I: Participants insert low FBN R/S ONP for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.

ARM II: Participants insert to low FBN > 99% S ONP product for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.

ARM III: Participants insert to high R/S ONP product for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.

ARM IV: Participants insert high FBN > 99% S ONP product for 4 weeks. Participants also attend 2 study visits and undergo oral mucosa sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Read and speak English
* At least 21 years old
* Willing to provide informed consent and abstain from all tobacco, nicotine, and marijuana use for at least 12 hours prior to Phase 1 study visits
* Willing to attend all study visits and use study ONPs
* Owns a smartphone and able to receive short messaging service (SMS) text messages with embedded survey link (for daily diary reports of ONP and other tobacco use)
* Negative pregnancy test produced during Phase 1 visits 1-5 and Phase 2 visit 1 if capable of becoming pregnant
* Exhaled carbon monoxide (CO) reading < 10 (Phase 1)
* CIGARETTE SMOKERS ONLY: Established cigarette smoker (has smoked at least 100 cigarettes, has smoked daily for at least the past 3 months, now smokes at least 5 cigarettes per day)
* ST USERS ONLY: Established moist snuff user (has used moist snuff daily for at least the past 3 months, uses at least 1.5 cans/week (as in Pickworth et al., 2014)

Exclusion Criteria:

* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress within the past 3 months
* Currently pregnant, planning to become pregnant, or breastfeeding (will be verified with urine pregnancy test before each Phase 1 study visit [acute use of usual product and study ONPs] and Phase 2 study visit 1 [distribution of study ONPs for outpatient ad libitum use])
* Currently engaging in tobacco quit attempt, interested in quitting all tobacco, or planning on quitting all tobacco in the next 3 months
* Oral or systemic health issues that affect oral microbiome or epithelium, including having fewer than 21 teeth, diabetes mellitus, or autoimmune disease (e.g., rheumatoid arthritis, lupus)
* CIGARETTE SMOKERS ONLY: Use of non-cigarette tobacco products ≥ 10 of the past 30 days
* CIGARETTE SMOKERS ONLY: Self-reported diagnosis of lung disease including asthma (if uncontrolled or worse than usual), cystic fibrosis, or chronic obstructive pulmonary disease
* CIGARETTE SMOKERS ONLY: Roll-your-own cigarette smokers
* ST USERS ONLY: Use of non-moist-snuff tobacco products ≥ 10 of the past 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Increased nicotine delivery | Up to 3 months
  Data will be used to assess the effects of nicotine concentration, form and isomer on the addiction potential and appeal of oral nicotine pouches (ONPs) relative to cigarettes and smokeless tobacco (ST). Generalized mixed effects models will be used to assess differences between the four ONP conditions and the usual product.
Liking | Up to 3 months
  Data will be used to assess the effects of nicotine concentration, form and isomer on the addiction potential and appeal of ONPs relative to cigarettes and ST. Generalized mixed effects models will be used to assess differences between the four ONP conditions and the usual product.
Craving/withdrawal suppression | Up to 3 months
  Data will be used to assess the effects of nicotine concentration, form and isomer on the addiction potential and appeal of ONPs relative to cigarettes and ST. Generalized mixed effects models will be used to assess differences between the four ONP conditions and the usual product.
Rate of switching to ONP | Up to 3 months
  Data will be used to assess the effects of nicotine concentration, form and isomer on the addiction potential and appeal of ONPs relative to cigarettes and ST. Generalized mixed effects models will be used to assess differences between the four ONP conditions and the usual product.
Rate of switching to ONPs | Up to 3 months
  Data will be used to evaluate the effects of nicotine concentration, form and isomer on switching from cigarettes or ST to ONPs either partially or completely. Logistic regression models will be used to examine whether differences in form and isomer significantly impact switching.

CONTACTS AND LOCATIONS:
Overall Officials: Brittney L Keller-Hamilton, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu